CLINICAL TRIAL: NCT02845115
Title: Pilot Study Evaluating Surgical Optimizing of a Middle Ear Implant (MET )With Laser Velocimetry in Patients With Moderate to Severe Hearing Loss in Case of Failure of Conventional Equipment
Brief Title: Surgical Optimizing of a Middle Ear Implant (MET )With Laser Velocimetry in Patients With Moderate to Severe Hearing Loss in Case of Failure of Conventional Equipment
Acronym: IOM laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2011.679
Record Dates: First submitted 2016-07-20; First posted 2016-07-27 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2016-07

CONDITIONS: Moderate to Severe Hearing Loss; Indication of Middle Ear Implant (MET)
Keywords: Middle Ear Implant; laser velocimetry

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (Other): standard care : usual technique for implanting
  Interventions: Device: Conventional implantation
- laser velocimetry (Experimental): optimized implantation of laser velocimetry
  Interventions: Device: optimized implantation with laser velocimetry

INTERVENTIONS:
Device: Conventional implantation — Usual implantation technique of a middle ear implant. The principle of the ossicular stimulator middle ear transducer MET 7000 (Middle Ear Transducer, METTM) is to directly transmit sounds on the ossicles bypassing the outer ear. Their constraint is the surgical placement of the implant.
  MET 7000 system (OTOLOGICS LLC, USA) is the implant that the investigators will use for their patients. The stimulator is usually placed against the body of the anvil by simple contact in the case of sensorineural hearing loss. In the case of mixed hearing loss, the stimulator will come in contact with the bracket using a titanium clip (ossicular prosthesis used in otologic surgery for ossiculoplasties). The optimized version corresponds to the use of the conventionally used in mixed deafness and applied to neurosensory deafness art. It is screwed onto the mastoid bone, the motor is suspended in the mastoid cavity and transmits vibrations to the body of the anvil by simple contact of the transducer.
  Arms: control
Device: optimized implantation with laser velocimetry
  Other Names: Group benefiting from the implantation technique optimized by laser velocimetry of a middle ear implant.( the MET ossicular stimulator 7000 the company "Otologics LLC")
  Arms: laser velocimetry

SUMMARY:
The aging of the population, and greater exposure to noise, are responsible for an increased incidence of hearing loss (presbycusis). This hearing loss is sensorineural disability that has become a real public health problem. The main means of rehabilitation of this disability is represented by the apparatus of patients with conventional hearing aids. However, these hearing aids have several drawbacks that limit their profits, often abandoning the prosthesis by the patient.

Middle ear implants were developed to answer these problems. They are intended to amplify the sound signal by transmitting directly to the middle ear to compensate for the hearing loss and are indicated in case of failure or contraindication of conventional equipment. However, these middle ear implants currently have limitations as performance failure. Recent data show that the performance of the ossicles repair techniques are dependent on the coupling of the ossicular prosthesis to the ossicles. Furthermore, advances in the understanding of the biomechanics of the ossicles confirm the importance of the placement and linkage of surgical restoration processes. This data can be applied to middle ear implants to improve performance. Indeed, a preliminary experimental study on anatomical parts, using analysis of the vibration of the middle ear structures by laser velocimetry, allowed the investigators to define the transducer placement method and coupling method to ossicles.

Investigators wish to validate in vivo results in a pilot study on a small number of patients by comparing two surgical techniques guided by velocimetric measures.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 60 years;
* Having given written informed consent prior to any procedure related to the study;
* Covered by a Health System where applicable, and/or in compliance with the recommendations of the national laws in force relating to biomedical research.
* Indication and IOM implantation request by the patient with a patient physically, psychologically and legally able to ask its implementation
* Average deafness to severe (mean thresholds between 40 to 90 dB) with speech discrimination> 40% to 75 dB.
* Deafness of pure perception or mixed hearing loss
* Non-fluctuating deafness over the last two years
* Failed or cons-indication to conventional equipment
* Rocky Scanner and MRI normal brain
* Patient fluent in French (to ensure validity audiological measures

Exclusion Criteria:

* Pregnant women or likely to be during the study.
* Not affiliated with a social security scheme Patients
* Major Patients protected by provisions of the law (Public Health Code).
* Refusal of consent.
* Ongoing Participation in another study that may interfere with the proposed study (investigator assessment).
* Existence of a cons-indication for surgery or port of the implant
* Motivation only aesthetic, evaluated by the principal investigator.
* Inability of predictable medium-term monitoring.
* Acoustic neuroma, tumors and other evolutionary processes of the rock and the cerebellopontine angle.
* Pathology requiring follow-up MRI (IOM against-indicating MRI).
* Patient with against-indication to MRI.
* Contraindication to the establishment of a pacemaker ossicular MET

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-02; Primary Completion 2015-02 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change from Baseline hearing at 8 months post-implantation (hearing gain), measured by tone and speech audiometry | at baseline (day 0) and 8 months
  The hearing will be measured by tone and speech audiometry in silence and in noise (dB) Results will be averaged per patient.

SECONDARY OUTCOMES:
Number of surgical implantation performed for the surgical laser velocimetry optimization technique | at 14 months
  number of surgical implantations performed in the required conditions and, if necessary, deviations will be described.
description of adverse events throughout the study | pre and post-operatively at day 0, at day 4, day 8 and then at 2, 3, 4, 5, 6, 7, 8 and 14 months.
Middle ear transfer function measured by laser velocimetry | pre-operatively at day 0 and then at 2, 3, 8 and 14 months.
  measured in mm/s/Pa
Tone and speech audiometry in silence and in noise (dB) | Baseline at inclusion visit, day 0, and then at 2, 3, 4, 5, 6, 7, 8 and 14 months.
Change in the quality of life measured by GHSI (Glasgow Health Status Inventory) score | day 0, and 2, 3, 5, 8 and 14 months.
  Changes will be described in both groups. GHSI questionnaire appreciate the impact of hearing loss on quality of life and whose translation is adapted to the French context.
Change in the quality of life measured by GBI (Glasgow Benefit Inventory) score | day 0, and 2, 3, 5, 8 and 14 months.
  Changes will be described in both groups. GBI questionnaire appreciate the benefit of the port of hearing aid before surgery and the benefit of the middle ear implant after the surgery.
Change in the quality of life measured by APHAB ( Abbreviated Profile of Hearing Aid Benefit) score | day 0, and 2, 3, 5, 8 and 14 months.
  Changes will be described in both groups. APHAB questionnaire is validated in subjects deaf to assess the discomfort associated with deafness in conditions of erveday life.
Change in the quality of life measured by SSQ (Speech Saptial Qualiteies) score | day 0, and 2, 3, 5, 8 and 14 months.
  Changes will be described in both groups. SSQ questionnaire evaluate the binaural hearing.